CLINICAL TRIAL: NCT02572609
Title: Relative Bioavailability Study Between Two Formulations Containing Ambroxol Hydrochloride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.509
Record Dates: First submitted 2015-10-05; First posted 2015-10-09 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

ARMS (2):
- Mucosolvan ® adult syrup (Experimental)
  Interventions: Drug: Mucosolvan ® adult syrup
- Ambroxol hydrochloride soft pastille (Experimental)
  Interventions: Drug: Ambroxol hydrochloride soft pastille

INTERVENTIONS:
Drug: Ambroxol hydrochloride soft pastille
  Arms: Ambroxol hydrochloride soft pastille
Drug: Mucosolvan ® adult syrup
  Arms: Mucosolvan ® adult syrup

SUMMARY:
to evaluate the bioavailability of ambroxol hydrochloride soft pastilles (test formulation), manufactured by Bolder Arzneimittel GmbH & Co. KG to Boehringer Ingelheim compared to ambroxol hydrochloride syrup (Mucosolvan® adult syrup), manufactured by Boehringer Ingelheim do Brasil Química e Farmacêutica Ltda.

ELIGIBILITY:
Inclusion criteria:

* The volunteer is between 18 and 50 years old, is a man or a woman who is not pregnant and/or in breastfeeding regime, and undertakes to use effective birth control method throughout the study period.
* Body mass index higher than or equal to 18.5 and lower than or equal to 29.9 kg/m2.
* The volunteer is in good health status and is with no clinically significant diseases, at the discretion of the physician as Medical History, measurements of Blood Pressure, Pulse and Temperature, Physical Examination, Electrocardiogram and complementary Laboratory Tests.
* Volunteer able to understand the nature and objective of the study, including the risks and adverse effects, with the intention to cooperate with the investigator and act in accordance with the requirements of the entire trial, which has to be confirmed by signing the Informed Consent Form.

Exclusion criteria:

* Volunteer has a known hypersensitivity to study drug or chemically related compounds; or to excipients described in adult syrup and/or soft pastille, for example, sorbitol (fructose).
* History or presence of gastrointestinal or liver diseases, or other condition that interferes with the absorption, distribution, excretion or metabolism of the drug.
* Use of maintenance therapy with any drug, except contraceptives.
* Diseases or health problems
* History of liver, renal, pulmonary, gastrointestinal, neurological, hematological, psychiatric, cardiac or allergic disease of any cause that requires pharmacological treatment or is considered to be clinically relevant by the investigator;
* Electrocardiographic findings not recommended, at the discretion of the investigator the participation in the study.
* Additional laboratory test results out of normal values according to the standard of this Potocol, unless they are considered clinically not significant by the investigator.
* Tabagism.
* Daily intake of more than 5 cups of coffee or tea.
* History of alcohol or drug abuse.
* Use of regular medication within 2 weeks prior to the initiation of this study, or use of any medication one week before starting this study.
* Hospitalization for any reason up to 8 weeks before starting the first treatment period of this study.
* Treatment within 3 months prior to this study treatment initiation with any drug that is known to have a well-defined toxic potential in large organs.
* Participation in any pharmacokinetic study with more than 300 mL of blood taken or ingested any - study drug within six months preceding the treatment start of this study.
* Donation or loss of 450 mL or more of blood within three months preceding the study or who donated more than 1500 mL within 12 months prior to this study treatment initiation.
* Pre-Confinement Examination Results
* Positive result for urine βHCG test carried out in female volunteers. Other conditions
* Any condition that prevents participation in the study as judged by the investigator.

Ages: 18 Years to 50 Years | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The crossover design 2x2 was used in the study. This is a conventional nonreplicated design with two formulations, two periods, two sequences (RT and TR) where each individual is randomly allocated in one of these sequences.
Groups:
- Sequence: TR: 01 pastille, single dose of Ambroxol hydrochloride soft pastille 15 mg (Test product) in period 1 and 2.5 mL, single dose, of Mucosolvan ® adult syrup (Reference product) in period 2.
  Washout period: 7 days
- Sequence: RT: 2.5 mL, single dose, of Mucosolvan ® adult syrup (Reference product) in period 1 and 01 pastille, single dose, of Ambroxol hydrochloride soft pastille 15 mg (Test product) in period 2.
  Washout period: 7 days
Period: Period 1: Treatment Period 1 + Washout
Arm/Group | Sequence: TR | Sequence: RT
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2: Treatment Period 2
Arm/Group | Sequence: TR | Sequence: RT
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): 36 subjects took 1 dose of reference product and 1 dose of test product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence: TR | Sequence: RT | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.39 (5.80) | 31.22 (7.30) | 30.30 (6.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: Maximum plasma concentration achieved
Time Frame: 0:00h (hours), 0:15h, 0:30h, 0:45h, 1:00h, 1:15h, 1:30h, 1:45h, 2:00h, 2:20h, 2:40, 3:00, 3:30h, 4:00h, 5:00h, 6:00h, 8:00h, 12:00h, 16:00h, 24:00h, 36:00h and 48:00h
Population: The pharmacokinetic set (PK Set): 36 subjects provided 1 evaluable value of reference product and 1 evaluable value of test product for the primary PK endpoints (Cmax and AUC0-t) without important protocol violations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Mucosolvan ® Adult Syrup: 2.5 mL, single dose, of Mucosolvan ® adult syrup 6 mg/mL (Reference product).
- Ambroxol Hydrochloride Soft Pastille: 01 pastille, single dose of Ambroxol hydrochloride soft pastille 15 mg (Test product).
Arm/Group | Mucosolvan ® Adult Syrup | Ambroxol Hydrochloride Soft Pastille
Number analyzed (Participants) | 18 | 18
ng/mL | 31.27 (30.38) | 35.50 (28.62)
Statistical Analysis 1: Comparison: Mucosolvan ® Adult Syrup vs Ambroxol Hydrochloride Soft Pastille; Test type: Non-Inferiority or Equivalence — Bioequivalence in the Cmax will be concluded if the 90% confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; p = 0.0082, Anderson-Hauck procedure; T/R Ratio = 113.56, 90% CI 2-sided [106.48 to 121.10], Standard Deviation 16.24 — Standard Deviation is actually the Coefficient of variation intra subject (CVintra)

2. Primary Outcome: AUC0-t
Description: Area under the plasma concentration-time curve, calculated by the trapezoidal methods from time 0 to time t, where t is the time for the last concentration experimentally determined above the Limit of Quantification (LOQ).
Time Frame: as for outcome 1
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Arm/Group | Mucosolvan ® Adult Syrup | Ambroxol Hydrochloride Soft Pastille
Number analyzed (Participants) | 18 | 18
ng.h/mL | 256.66 (33.36) | 307.00 (28.97)
Statistical Analysis 1: Comparison: Mucosolvan ® Adult Syrup vs Ambroxol Hydrochloride Soft Pastille; Test type: Non-Inferiority or Equivalence — Bioequivalence in the AUC0-t will be concluded if the 90% confidence interval for the test/reference ratio of the least squares means is fully contained within the acceptance range, 80.00% - 125.00%; p = 0.0438, Anderson-Hauck procedure; T/R Ratio = 119.61, 90% CI 2-sided [114.65 to 124.79], Standard Deviation 10.65 — Standard Deviation is actually the Coefficient of variation intra subject (CVintra)

ADVERSE EVENTS:
Time Frame: From first drug administration until 48 hours after last drug administration, upto 08 days
Arm/Group | Mucosolvan® Adult Syrup | Ambroxol Hydrochloride Soft Pastille
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.